CLINICAL TRIAL: NCT05804994
Title: A Randomized, Comparative Study to Evaluate the Efficacy and Tolerance of the Medical Device Elgydium Clinic Sensileave Gel (V063B - DP3003) on Dentin Hypersensitivity During Teeth Whitening.
Brief Title: Evaluate the Efficacy and the Tolerance of the Medical Device V063B-DP3003 on Dentin Hypersensitivity During Teeth Whitening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: V063B20220080
Record Dates: First submitted 2023-03-10; First posted 2023-04-07 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Tooth Whitening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical device group (Experimental): Group applying the tested medical device
  Interventions: Device: Elgydium Clinic Sensileave Gel (V063B - DP3003)
- Control group (No Intervention): Group not applying the tested medical device

INTERVENTIONS:
Device: Elgydium Clinic Sensileave Gel (V063B - DP3003) — Tested product is applied/used only once a day before whitening tray wear.
  Arms: Medical device group

SUMMARY:
A dental gel intended to relieve pain related to dentin hyper sensitivity is commercialized in several countries worlwide since May 2017. Its efficacy and tolerance has already been proven in dentin hyper sensitivity. In this new study, we assess the efficacy and tolerance of this tested product in a specific external agression, the teeth whitening.

DETAILED DESCRIPTION:
Comparative open-label PMCF (Post-Market Clinical Follow-up) randomized controlled study will be conducted as multicentric trial in adult with dentin hypersensitivity during their teeth whitening. To evaluate the efficacy and tolerance of the medical device Elgydium Clinic Sensileave Gel (V063B - DP3003) on dentin hypersensitivity during teeth whitening

4 visits are planned:

* Visit 1 (V1) - Selection
* Visit 2 (V2) - Start of teeth whitening
* Visit 3 (V3) - Start of tested product application - Inclusion / Randomization
* Visit 4 (V4) - Study end

ELIGIBILITY:
Inclusion Criteria:

* Subject who has a pain score (i.e. maximum intensity felt while the whitening tray wear) of at least 3 on a NRS ranging from 0 (None) to 10 (Severe) evaluated since the beginning of his teeth whitening.
* Subject wishing to have a teeth whitening
* Subject with a healthy gum status according to the investigator
* Subject with at least 20 natural teeth

Exclusion Criteria:

Related to the teeth condition:

* Subject with active teeth decay
* Subject with teeth showing evidence of facets of attrition, premature contact, cracked enamel on the teeth to be studied and adjacent teeth
* Subject with teeth showing evidence of irreversible pulpitis and active periodontal disease
* Subject having a cutaneous-mucosal disease liable to interfere with study data according to the investigator
* Subject with an odontological condition, an acute chronic or progressive disease or history of disease considered by the investigator hazardous for the subject or incompatible with the study

Related to the treatment/product:

* Subject having undergone professional desensitizing therapy in the mouth
* Systemic treatment/product and topical treatment/product in the mouth liable to interfere with study data according to the investigator assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the soothing effect of the medical device Elgydium Clinic Sensileave Gel (V063B - DP3003) on dentin hypersensitivity due to teeth whitening | About 10 days
  NRS ranging from 0 (None) to 10 (Severe)

SECONDARY OUTCOMES:
Evaluate the soothing effect of the medical device Elgydium Clinic Sensileave Gel (V063B - DP3003) on dentin hypersensitivity due to teeth whitening | About 10 days
  The global duration (in hours) of wearing the whitening tray
Evaluate the soothing effect of the medical device Elgydium Clinic Sensileave Gel (V063B - DP3003) on dentin hypersensitivity due to teeth whitening | About 10 days
  Percentage of subjects who stopped at least once trays wear because of pain
Evaluate the soothing effect of the medical device Elgydium Clinic Sensileave Gel (V063B - DP3003) on dentin hypersensitivity due to teeth whitening | About 10 days
  The total number of days of not wearing trays due to pain
Evaluate the effect of the medical device Elgydium Clinic Sensileave Gel (V063B - DP3003) on teeth whitening | About 10 days
  Teeth colours evaluated by using VITA shades guides (Ranging from 1 to 16. Higher scores means a worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Dermscan Poland, Gdansk, Poland